CLINICAL TRIAL: NCT01059851
Title: An Open-Label, Single-Dose Study to Investigate the Pharmacokinetics of MK-4305 in Patients With Impaired Renal Function
Brief Title: Pharmacokinetics of Suvorexant in Participants With Impaired Renal Function (MK-4305-023)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4305-023; 2010_505 (Other: Merck Registration Number)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Participants with Severe Renal Impairment (Part I) (Experimental): Participants with severe renal impairment will receive a
  single dose of 20 mg open-label suvorexant during Part I of the
  study.
  Interventions: Drug: Suvorexant
- Healthy Participants (Severe Impairment Controls) (Part I) (Experimental): Healthy participants matched to participants with severe renal impairment will receive a single dose of 20 mg open-label suvorexant during Part I of the study.
  Interventions: Drug: Suvorexant
- Participants with Moderate Renal Impairment (Part II) (Experimental): Participants with moderate renal impairment will receive a single dose of 20 mg open-label suvorexant during Part II of the study.
  Interventions: Drug: Suvorexant
- Healthy Participants (Moderate Impairment Controls) (Part II) (Experimental): Healthy participants matched to participants with moderate renal impairment will receive a single dose of 20 mg open-label suvorexant during Part II of the study.
  Interventions: Drug: Suvorexant
- Participants with Mild Renal Impairment (Part II) (Experimental): Participants with mild renal impairment will receive a single dose of 20 mg open-label suvorexant during Part II of the study.
  Interventions: Drug: Suvorexant
- Healthy Participants (Mild Impairment Controls) (Part II) (Experimental): Healthy participants matched to participants with mild renal impairment will receive a single dose of 20 mg open-label suvorexant during Part II of the study.
  Interventions: Drug: Suvorexant

INTERVENTIONS:
Drug: Suvorexant — single oral dose of 20 mg (administered as 2 x 10 mg tablets) of suvorexant administered with ~240 mL of water after an 8 hour fast
  Other Names: MK-4305

SUMMARY:
This study will investigate whether the plasma concentration-time profile and pharmacokinetics (PK) of suvorexant (MK-4305) in participants with impaired renal function are similar to those observed in healthy participants; and will evaluate the safety and tolerability of suvorexant both in participants with impaired renal function and in healthy participants.

DETAILED DESCRIPTION:
Study Design:

This study plans to enroll 16 participants in Part I (8 participants with severe renal impairment and a control group of 8 healthy participants) and 32 participants in Part II (8 participants with moderate renal impairment and a control group of 8 healthy participants; and 8 participants with mild renal impairment and a control group of 8 healthy participants).

Part II will be conducted only if the primary hypothesis is not met in Part I and there is a significant difference in the PK of suvorexant between healthy participants and severe renal impairment participants.

ELIGIBILITY:
Inclusion Criteria:

Impaired Renal Function Participants:

* Females of reproductive potential must have a negative pregnancy test and agree to use (and/or have their partner use) two acceptable methods of birth control
* Body Mass Index (BMI) ≤40 kg/m^2
* Diagnosis of renal insufficiency

Healthy Participants:

* Females of reproductive potential must have a negative pregnancy test and agree to use (and/or have their partner use) two acceptable methods of birth control
* Body Mass Index (BMI) ≤40 kg/m^2 and is matched for BMI ± 5 units to his/her corresponding renal participant
* In general good health
* Matched for age ± 10 years to his/her corresponding renal participant

Exclusion Criteria:

Impaired Renal Function Participants:

* Is mentally or legally incapacitated
* History of a clinically significant psychiatric disorder over the last year
* Has rapidly fluctuating renal function or has demonstrated or suspected renal artery stenosis
* Has had a kidney transplant
* Unstable endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary diseases
* History of cancer (Some exceptions apply)
* Regular user of barbiturates or sleep aides
* Consumes excessive amounts of alcohol (>2 drinks/day)
* Consumes excessive amounts of caffeinated beverages (>6/day)
* Has had major surgery within 4 weeks
* Has a history of significant multiple and/or severe allergies
* Has a history of cataplexy
* Participant works a night shift and is not able to avoid night shift work during the study
* Current or history of illicit drug abuse
* Nursing mothers

Healthy Participants:

* Is mentally or legally incapacitated;
* Has a history of stroke, chronic seizures, or major neurological disorder
* Unstable endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary diseases
* History of cancer (Some exceptions apply)
* Regular user of barbiturates or sleep aides
* Consumes excessive amounts of alcohol (>2 drinks/day)
* Consumes excessive amounts of caffeinated beverages (>6/day)
* Has had major surgery within 4 weeks
* Has a history of significant multiple and/or severe allergies
* Has a history of cataplexy
* Participant works a night shift and is not able to avoid night shift work during the study
* Current or history of illicit drug abuse
* Nursing mothers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05-24 (Actual); Primary Completion 2010-07-15 (Actual); Study Completion 2010-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-023&kw=4305-023&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were enrolled in Part I of the study. Because the primary hypothesis was met in Part I, no participants were enrolled in Part II of the study.
Groups:
- Participants With Severe Renal Impairment (Part I): Participants with severe renal impairment received a
  single dose of 20 mg open-label suvorexant.
- Healthy Participants (Severe Impairment Controls) (Part I): Healthy participants matched to participants with severe renal impairment received a single dose of 20 mg open-label suvorexant.
- Participants With Moderate Renal Impairment (Part II): Participants with moderate renal impairment were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled in this arm.
- Healthy Participants (Moderate Impairment Controls) (Part II): Healthy participants matched to participants with moderate renal impairment were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled in this arm.
- Participants With Mild Renal Impairment (Part II): Participants with mild renal impairment were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled in this arm.
- Healthy Participants (Mild Impairment Controls) (Part II): Healthy participants matched to participants with mild renal impairment were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled in this arm.
Period: Overall Study
Arm/Group | Participants With Severe Renal Impairment (Part I) | Healthy Participants (Severe Impairment Controls) (Part I) | Participants With Moderate Renal Impairment (Part II) | Healthy Participants (Moderate Impairment Controls) (Part II) | Participants With Mild Renal Impairment (Part II) | Healthy Participants (Mild Impairment Controls) (Part II)
Started | 8 | 8 | 0 | 0 | 0 | 0
Completed | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only presented for participants in Part I of the study (N=16). No participants were enrolled in Part II of the study.
Groups:
- Healthy Participants (Part I): Healthy participants matched to participants with severe renal impairment received a single dose of 20 mg open-label suvorexant.
- Total: Total of all reporting groups
Arm/Group | Participants With Severe Renal Impairment (Part I) | Healthy Participants (Part I) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.5) | 48.1 (11.6) | 49.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to Infinity (0-∞) After Single Dose Suvorexant: Severe Renal Impairment Participants Versus Healthy Participants (Part I)
Description: Overall exposure was assessed by the area under the plasma concentration versus time curve from time zero to infinity (AUC[0-∞]). AUC(0-∞) was calculated as the sum of the AUC to the last time point with a detectable plasma concentration (AUC[0-last]) and the extrapolated area given by the quotient of the last detectable concentration and the apparent terminal rate constant (λ).
Time Frame: Predose and 0.5, 1, 2, 4, 6, 9, 12, 16, 24, 48, 72, 96, and 120 hours post-dose
Population: All Treated Participants
Measure: Geometric Mean (95% Confidence Interval); unit: μM•hr
Arm/Group | Participants With Severe Renal Impairment (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
μM•hr | 11.98 [9.45 to 15.20] | 9.81 [7.72 to 12.47]
Statistical Analysis 1: Comparison: Participants With Severe Renal Impairment (Part I) vs Healthy Participants (Part I); The geometric mean (GM) for each participant group and the corresponding 95% confidence interval (CI) were calculated for AUC(0-∞) using an analysis of covariance (ANCOVA) model. The AUC(0-∞) geometric mean ratio (GMR) of the 2 participant groups was used to test the primary hypothesis, which was that the AUC(0-∞) of suvorexant following a single oral dose would be similar between participants with renal impairment and healthy matched control participants; Test type: Non-Inferiority or Equivalence — AUC(0-∞) GMR = AUC(0-∞) GM for Severe Renal Impairment Participants ÷ AUC(0-∞) GM for Healthy Participants. A 90% CI for the AUC(0-∞) GMR was computed from the ANCOVA model. As prespecified by the analysis plan, if the 90% CI for the AUC(0-∞) GMR was contained within the interval [0.50, 2.00], then the hypothesis would be met and the AUC(0-∞) of suvorexant would be similar in both groups of participants. That is, if the true ratio of the GM AUC(0-∞) is greater than 0.50 and no more than 2.00; ANCOVA; AUC(0-∞) Geometric Mean Ratio = 1.22, 90% CI 2-sided [0.93 to 1.60]

2. Primary Outcome: AUC(0-∞) After Single Dose Suvorexant: Moderate and Mild Renal Impairment Participants Versus Healthy Participants (Part II)
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 4, 6, 9, 12, 16, 24, 48, 72, 96, and 120 hours post-dose
Population: Per protocol, the decision to conduct Part II of study in moderate/mild renal impairment participants was conditional on results of AUC (0-∞) analysis in severe renal impairment participants (Part I). Based on results of Part I of study, Part II was not conducted and AUC(0-∞) analysis in moderate/mild renal impairment was not done.
Arm/Group | Participants With Moderate Renal Impairment (Part II) | Healthy Participants (Moderate Impairment Controls) (Part II) | Participants With Mild Renal Impairment (Part II) | Healthy Participants (Mild Impairment Controls) (Part II)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug.
Time Frame: From administration of study drug through 14 days after administration of study drug
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Participants With Severe Renal Impairment (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
participants | 2 | 4

4. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 3
Time Frame: From administration of study drug through 14 days after administration of study drug
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Participants With Severe Renal Impairment (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From administration of study drug through 14 days after administration of study drug
Arm/Group | Participants With Severe Renal Impairment (Part I) | Healthy Participants (Part I)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Severe Renal Impairment (Part I) (N=8) | Healthy Participants (Part I) (N=8)
dry mouth (Gastrointestinal disorders) | 0 | 2
headache (Nervous system disorders) | 0 | 3
somnolence (Nervous system disorders) | 1 | 0
oligomenorrhoea (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.